CLINICAL TRIAL: NCT02867917
Title: Comparison of Taste and Texture of Metamucil, Volcolon and Psyllium Orange Generic
Brief Title: Comparison of Taste and Palatability in Fiber Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, PF Vollebregt, MD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 2016.360
Record Dates: First submitted 2016-08-10; First posted 2016-08-16 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Constipation
Keywords: Fibers; Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Total group (Other): Volcolon sugar free & Metamucil Orange & Psyllium Orange in a randomized order.
  Interventions: Drug: Volcolon sugar free; Drug: Metamucil Orange; Drug: Psyllium Orange

INTERVENTIONS:
Drug: Volcolon sugar free — 1 sachet contains 4 g powder 980mg/g psyllium fibers x 4 g per sachet = 3.92 g psyllium fibers/sachet
Drug: Metamucil Orange — 1 sachet contains 3.4 g psyllium fibers So 25 ml contains 0.425 g psyllium fibers
Drug: Psyllium Orange — 1 sachet contains 3.25 g psyllium fibers So 25 ml contains 0.406 g psyllium fibers

SUMMARY:
The purpose of this study is to compare 1. taste and 2. texture/palatability of Metamucil orange®, Volcolon® and generic orange psyllium.

DETAILED DESCRIPTION:
Background of the study:

A pleasant taste of a prescription improves patient compliance and adherence. According to the literature, only 50% of patients who suffer from chronic diseases adhere to treatment recommendations (1). This results in suboptimal outcomes (2). There are numerous factors that affect adherence, including characteristics of the illness, interaction between physician and patient, the complexity and duration of treatment, side effects of treatment and costs of treatment (3). Furthermore, medication palatability is also crucial for adherence. Several studies have addressed the palatability of medication for different disorders, like hypertension, HIV and Alzheimer's disease (4-6). Therefore, pharmaceutical companies pay attention to manufacture more formulations and add pleasant flavours which may improve the palatability. Fiber supplements are increasingly used for treatment of chronic constipation both in adults and children. In the Netherlands several formulas are available such as Metamucil orange®, Volcolon® en generic psyllium orange. These are effective and save formulas. Little literature is available concerning taste and laxatives or fibers, although many patients complain about taste and texture of the preparations. Studies with polyethylene glycol preparations performed by our research group demonstrated some differences in palatability between these preparations (7-9). There are hardly any studies about fibers and taste. The taste is mentioned to be acceptable; one study compares dried prunes with psyllium and concludes there is no difference in taste experience (10). In order to improve patient compliance, it is of clinical importance to know which preparations are the most acceptable to the patient, and use that as first choice. We hypothese that the taste and palatability of Metamucil orange® is preferable.

Objective of the study:

Comparison of 1. taste and 2. texture/palatability of Metamucil orange®, Volcolon® and generic orange psyllium.

Study design:

It is a double blind, randomized, crossover study.

Study population:

100 healthy volunteers (primary recruitment of medical students).

Intervention: All healthy volunteers will try the 3 different formulas. After swallowing the first formula, the mouth will be rinsed with water. Then the second formula will be tried, after rinsing the mouth again the third formula will be tried. Every time after tasting a formula, the questionnaire is filled in, before starting with the next formula. The maximum intake is 3 x 25 ml (75 ml), this is 37,5% of one dosage advised quantity of fibre. The sequence in which the formulas are tasted is randomized.

Preparations and dosage

Each sachet needs to be solved in a glass of water. This matches (approximately) 200 ml. During the study the volunteers will taste 3 x 25 ml of water. This matches 37,5% of one dosage. The average intake of psyllium fibers is 1-3 sachets a day. Dosage if the different products:

* Volcolon sugar free (Dutch name: Volcolcolon suikervrij): 1 sachet contains 4 g powder o 980mg/g psyllium fibers x 4 g per sachet = 3.92 g psyllium fibers/sachet o So 25 ml contains 0.490 g psyllium fibers
* Metamucil Orange: 1 sachet contains 3.4 g psyllium fibers o So 25 ml contains 0.425 g psyllium fibers
* Psyllium Orange: 1 sachet contains 3.25 g psyllium fibers o So 25 ml contains 0.406 g psyllium fibers These three products are the most used products for each brand (Metamucil orange, Volcolon and generic orange). This leads to the greatest coverage of the three brands in the Netherlands. The volunteers will swallow 25 ml of each product, three in total. This leads to an intake of 1.32 g (0.490 g + 0.425 g + 0.406= 1.32 g) psyllium fibers.

According to the Dutch Board of Health (in Dutch: Gezondheidsraad) the average intake of fibers should be between 30 and 40 g a day. So, the volunteers will swallow approximately 4% (3.3 - 4.4%) of the advised intake of fibers. Therefore, we do not expect any problems when the volunteers swallow these products.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness (if applicable): The maximum intake is 3 x 25 ml (75 ml), this is 37,5% of one dosage advised quantity of fibre. Therefore, we do not expect any problems when the volunteers swallow these products.

References:

1. World Health Organisation. Adherence to long term therapies: evidence for action. 2003.
2. Osterberg L, Blaschke T. Adherence to medication 1. N Engl J Med 2005 August 4;353(5):487-97.
3. Ingersoll KS, Cohen J. The impact of medication regimen factors on adherence to chronic treatment: a review of literature 1. J Behav Med 2008 June;31(3):213-24.
4. Van der Linden D, Callens S, Brichard B, Colebunders R. Pediatric HIV: new opportunities to treat children 1. Expert Opin Pharmacother 2009 August;10(11):1783-91.
5. Meier CM, Simonetti GD, Ghiglia S, Fossali E, Salice P, Limoni C et al. Palatability of angiotensin II antagonists among nephropathic children 1. Br J Clin Pharmacol 2007 May;63(5):628-31.
6. Yan YD, Woo JS, Kang JH, Yong CS, Choi HG. Preparation and evaluation of taste-masked donepezil hydrochloride orally disintegrating tablets 1. Biol Pharm Bull 2010;33(8):1364-70.
7. Felt-Bersma R.J., Kooyman G., Kuipers E.J. Colonic lavage prior to colonoscopy: comparable outcomes of two polyethylene-glycol preparations and a sodium-phosphate solution. Ned Tijdschr Geneeskd. 2004 Jan 24; 148 (4): 181-5
8. Szojda MM, Mulder CJ, Felt-Bersma RJ. Differences in taste between two polyethylene glycol preparations.J Gastrointestin Liver Dis. 2007;16(4):379-81
9. Lam TJ, Mulder CJ, Felt-Bersma RJ. Differences in taste between three polyethylene glycol preparations: a randomized double-blind study. Patient Prefer Adherence. 2011;5:423-6.
10. Yan YD, Woo JS, Kang JH, Yong CS, Choi HG. Preparation and evaluation of taste-masked donepezil hydrochloride orally disintegrating tablets 1. Biol Pharm Bull 2010;33(8):1364-70.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* In good health
* Able to understand the instruction and give informed consent

Exclusion Criteria:

* Gastrointestinal problems
* Swallowing disorders
* Rheumatic related diseases
* Known hypersensitivity to the study medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Taste: 5-point likert scale | Directly after consuming the fiber (1 minute)
  1. = very poor taste / unpleasant
  2. = poor taste / unpleasant
  3. = neutral
  4. = tasty / pleasant
  5. = very tasty/ very pleasant
Texture: 5-point likert scale | Directly after consuming the fiber (1 minute)
  1. = very poor taste / unpleasant
  2. = poor taste / unpleasant
  3. = neutral
  4. = tasty / pleasant
  5. = very tasty/ very pleasant

CONTACTS AND LOCATIONS:
Overall Officials: Richelle JF Felt-Bersma, MD, PhD, Principal Investigator — VU Medical Center Amsterdam

IPD SHARING:
Plan to Share IPD: No